CLINICAL TRIAL: NCT00979056
Title: Prospective, Randomised, Placebo Controlled, Double Blind Monocenter Trial for the Prophylactic Treatment of Diarrhoea With Rifaximin for Travellers to South- and Southeast-Asia
Brief Title: Prophylactic Treatment of Travellers' Diarrhoea With Rifaximin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Philipp Zanger, MD MSc DTM (Other)
Responsible Party: Sponsor-Investigator, Dr. Philipp Zanger, MD MSc DTM, Oberarzt, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Rifa1; 2007-003986-42
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Diarrhoea
Keywords: Traveller's diarrhoea; Prevention
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Lactose (Placebo Comparator)
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: Rifaximin — 400 mg per day, oral use, maximum duration 28 days
  Other Names: Xifaxan; Normix; ATC code A07AA11; Chemical Abstracts Service (CAS) 80621814
  Arms: Rifaximin
Drug: Lactose — Coated Tablet, Oral Use
  Arms: Lactose

SUMMARY:
The aim of the study is to investigate the efficacy of the prophylactic treatment with rifaximin to prevent travellers diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 and < 65 years
* Good general condition (according to history and clinical examination)
* Written informed consent
* No pregnancy
* No breast feeding
* Efficacious contraception (e.g. oral, double-barrier) during the study and 4 weeks after termination of the study
* No participation in other clinical trials 4 weeks before, during participation, and 4 weeks after participation in this study
* Planned travel period between 6 and 28 days
* Planned travel to South- and Southeast Asia
* Planned time to arrival in South- or Southeast Asia ≤ 24 hours

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Age < 18 and ≥ 65 years
* No written informed consent
* Chronic gastrointestinal disease and/ or immune insufficiency
* Low general condition (according to history and clinical examination)
* Regular medication with gastrointestinal side-effects and/or immunosuppressive medication
* Participation in other clinical trials 4 weeks before, during and 4 weeks after termination of the study
* No efficacious contraception
* Planned travel period < 6 and > 28 days
* Planned travel outside South- and Southeast Asia
* Vaccination against cholera using DUKORAL within 12 months prior to inclusion
* Planned time to arrival in South- or Southeast Asia > 24 hours
* Known hypersensitivity against rifaximin or rifamycin-derivatives in general
* Known lactose intolerance

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of the prevention of travellers diarrhea with rifaximin by measurement of frequency and consistence of the stool. Diarrhea will be defined as passage of >2 unformed stools/24 hr plus one or more signs or symptoms of enteric infection. | From the first day of the travel (travel period between 6 and 28 days) to 1 week after the subject's return to Germany

SECONDARY OUTCOMES:
Documentation of adverse effects and tolerance of prophylaxis with rifaximin. | From the first day of the travel (travel period between 6 and 28 days) to 1 week after the subject's return to Germany
Evaluation of prevention of post infectious irritable bowel syndrome. | From the first day of the travel (travel period between 6 and 28 days) to 6 months after the subject's return to Germany

CONTACTS AND LOCATIONS:
Overall Officials: Philipp G. Zanger, MD MSc DTM, Principal Investigator — Institute of Tropical Medicine, University Hospital of Tübingen
Locations (1):
- Institute of Tropical Medicine, University Hospital of Tübingen, Tübingen, Germany

REFERENCES:
- [Result] Zanger P, Nurjadi D, Gabor J, Gaile M, Kremsner PG. Effectiveness of rifaximin in prevention of diarrhoea in individuals travelling to south and southeast Asia: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2013 Nov;13(11):946-54. doi: 10.1016/S1473-3099(13)70221-4. Epub 2013 Sep 4. PMID 24012319